CLINICAL TRIAL: NCT00475306
Title: A Randomized, Facorial Design Study to Optimize the Dose of Parenteral Metoclopramide
Brief Title: The Montefiore Metoclopramide Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Friedman, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-01-005
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-11

CONDITIONS: Nausea; Extrapyramidal Symptoms
Keywords: Metoclopramide; Nausea; Akathisia; Emergency department
MeSH Terms: conditions — Nausea; Psychomotor Agitation; Emergencies | interventions — Metoclopramide; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metoclopramide 20+diphenhydramine (Active Comparator): Metoclopramide 20 mg + diphenhydramine, delivered intravenously over 15 minutes
  Interventions: Drug: Diphenhydramine 25 mg; Drug: Metoclopramide 20 mg
- Metoclopramide 20+placebo (Active Comparator): Metoclopramide 20 mg + placebo, delivered intravenously over 15 minutes
  Interventions: Drug: Placebo; Drug: Metoclopramide 20 mg
- Metoclopramide 10 + placebo (Active Comparator): Metoclopramide 10mg + placebo, delivered intravenously over 15 minutes
  Interventions: Drug: metoclopramide 10 mg; Drug: Placebo
- Metoclopramide 10+diphenhydramine (Active Comparator): Metoclopramide 10 mg + diphenhydramine 25 mg, delivered intravenously over 15 minutes
  Interventions: Drug: metoclopramide 10 mg; Drug: Diphenhydramine 25 mg

INTERVENTIONS:
Drug: metoclopramide 10 mg — an anti-emetic medication
  Arms: Metoclopramide 10 + placebo; Metoclopramide 10+diphenhydramine
Drug: Diphenhydramine 25 mg — used for prophylaxis against akathisia
  Arms: Metoclopramide 10+diphenhydramine; Metoclopramide 20+diphenhydramine
Drug: Placebo — placebo
  Arms: Metoclopramide 10 + placebo; Metoclopramide 20+placebo
Drug: Metoclopramide 20 mg — Metoclopramide 20 mg
  Arms: Metoclopramide 20+diphenhydramine; Metoclopramide 20+placebo

SUMMARY:
Metoclopramide is a dopamine antagonist frequently used for the treatment of nausea, vomiting, and migraine headaches in Emergency Departments. However, little research has focused on the optimal dose of metoclopramide for treatment of nausea in the emergency department. We propose a randomized, double-blind, placebo controlled trial to investigate the optimal dose of metoclopramide for treatment of nausea.

DETAILED DESCRIPTION:
The most effective dose of metoclopramide for treatment of nausea in the emergency department setting has not been thoroughly investigated. One pilot study among emergency department patients in Australia found no statistical difference between 10 mg and 0.4 milligrams/kilogram; another investigation suggests that the anti-emetic effect of 10 milligrams of metoclopramide is no more effective than placebo. In contrast, investigations focusing on chemotherapy patients and post-operative patients suggest that higher dosage metoclopramide is more effective in treating nausea and vomiting. This emergency department study will compare the anti-emetic efficacy of 10 milligrams and 20 milligrams of metoclopramide by using the visual analog scale.

In addition to evaluation of dose, we will evaluate one of the most common side affects of metoclopramide, akathisia. Akathisia is characterized by a subjective component of restlessness and an objective component in the form of the inability to remain motionless. Anti-cholinergic medications are known to reduce extrapyramidal symptoms such as akathisia when dopamine function is impaired in the basal ganglia. In fact, the use of diphenhydramine has been shown to reduce the incidence of akathisia in patients receiving a different anti-emetic, prochlorperazine. However, no research has focused on the use of anti-cholinergic medications to reduce metoclopramide induced akathisia. This investigation will assess the use of 25 mg of diphenhydramine in preventing metoclopramide induced akathisia in ED patients being treated for nausea/vomiting.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary complaints of nausea/vomiting
* age 21-65

Exclusion Criteria:

* pregnancy
* use of anti-histamine or dopamine antagonist as outpatient and/or within last 24 hours of presentation
* previous adverse reaction to study medications
* use of opioid medications prior to study start time within that ED visit

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, Principal Investigator — Montefiore Medical Center; Brooke Bender, MD, Study Director — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who presented to one ED with nausea were eligible for participation
Groups:
- Metoclopramide 20 mg+Diphenhydramine: Metoclopramide 20mg co-administered with diphenhydramine 25 mg, intravenously
- Metoclopramide 20+Placebo: Metoclopramide 20 mg co-administered with placebo, intravenously
- Metoclopramide 10 + Placebo: Metoclopramide 10 mg co-administered with placebo, intravenously
- Metoclopramide 10+Diphenhydramine: Metoclopramide 10 mg co-administered with diphenhydramine 25 mg, intravenously
Period: Overall Study
Arm/Group | Metoclopramide 20 mg+Diphenhydramine | Metoclopramide 20+Placebo | Metoclopramide 10 + Placebo | Metoclopramide 10+Diphenhydramine
Started | 73 | 72 | 72 | 72
Completed | 72 (1 patient had resolution of nausea prior and did not receive the investigational medication) | 71 (For 1 patient, data collection was incomplete and results could not be analyzed) | 72 | 71 (1 patient's intravenous line infiltrated.)
Not Completed | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Metoclopramide 20mg+Diphenhydramine: Metoclopramide 20 mg co-administered with diphenhydramine 25mg, intravenously
- Metoclopramide 10+Diphenhydramine: Metoclopramide 10mg co-administered with diphenhydramine 25mg, intravenously
- Total: Total of all reporting groups
Arm/Group | Metoclopramide 20mg+Diphenhydramine | Metoclopramide 20+Placebo | Metoclopramide 10 + Placebo | Metoclopramide 10+Diphenhydramine | Total
Number analyzed (Participants) | 72 | 71 | 72 | 71 | 286
Age Continuous [Mean (Standard Deviation); unit: Years] | 39 (12) | 42 (14) | 40 (13) | 39 (13) | 40 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Please note: Only patients who completed the study are reported here
  Participants
    Female | 52 | 52 | 55 | 51 | 210
    Male | 20 | 19 | 17 | 20 | 76

OUTCOME MEASURES:

1. Primary Outcome: Nausea Scale
Description: Patients were asked to report their level of nausea on a scale for 0 to 10, with 0 representing no nausea and 10 the worst nausea imaginable
Time Frame: 60 minutes
Population: Only patients who received the investigational medication are included in this analysis. Please see the participant flow section for more details.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Metoclopramide 20mg+Diphenhydramine | Metoclopramide 20+Placebo | Metoclopramide 10 + Placebo | Metoclopramide 10+Diphenhydramine
Number analyzed (Participants) | 72 | 71 | 72 | 71
units on a scale | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]

2. Secondary Outcome: Number of Participants With Akathisia
Description: The akathisia outcome was reported as follows: Either development of akathisia as measured using the Short Akathisia Instrument (Vinson DR. Journal of Emergency Medicine. 2006; 31:139-145)or use of rescue medication for treatment of akathisia.The short akathisia instrument briefly measures subjective and objective restlessness.
Time Frame: 60 minutes
Population: Only patients who received the investigational medication are included in this analysis. Please see participant flow for details
Measure: Number; unit: participants
Arm/Group | Metoclopramide 20mg+Diphenhydramine | Metoclopramide 20+Placebo | Metoclopramide 10 + Placebo | Metoclopramide 10+Diphenhydramine
Number analyzed (Participants) | 72 | 71 | 72 | 71
participants | 9 | 12 | 5 | 8

ADVERSE EVENTS:
Arm/Group | Metoclopramide 20mg+Diphenhydramine | Metoclopramide 20+Placebo | Metoclopramide 10 + Placebo | Metoclopramide 10+Diphenhydramine
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/71 | 0/72 | 0/71
Other Adverse Events (participants affected / at risk) | 0/72 | 0/71 | 0/72 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes